CLINICAL TRIAL: NCT03748069
Title: Unraveling the Pathogenesis of Influenza-associated Aspergillosis: a Single-center, Prospective Cohort Pilot Study
Brief Title: Influenza Associated Aspergillosis In-depth Investigation
Acronym: PIAS
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: PIAS
Record Dates: First submitted 2018-10-04; First posted 2018-11-20 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-10

CONDITIONS: Influenza With Pneumonia; Invasive Pulmonary Aspergillosis
Keywords: Influenza; IPA; ICU; Immunology
MeSH Terms: conditions — Invasive Pulmonary Aspergillosis; Influenza, Human

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood, serum, white cells, broncho-alveolar lavage fluid, lung tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Influenza positive CAPIV: All consecutive patients older than 18 years, admitted to the ICU with respiratory distress with microbiologically confirmed diagnosis of influenza
- Influenza negative CAPIV: All consecutive patients older than 18 years, admitted to the ICU for respiratory distress due to community-acquired pneumonia (CAP) and with a microbiologically confirmed absence of influenza

SUMMARY:
This trial is aimed to study the immunological and pathological characteristics of influenza versus non-influenza severe community-acquired pneumonia patients in ICU.

DETAILED DESCRIPTION:
This trial is aimed to study the immunological and pathological characteristics of influenza versus non-influenza severe community-acquired pneumonia patients in ICU, and correlate findings with occurrence of secondary invasive pulmonary aspergillosis infection.

All consecutive patients aged 18 or older admitted to ICU during the inclusion period with respiratory distress due to influenza positive/negative community acquired pneumonia (CAP) will be included.

ELIGIBILITY:
Inclusion Criteria:

* All patients older than 18 years, admitted to ICU with respiratory distress with microbiologically confirmed diagnosis of influenza (for inclusion in the influenza group)
* All patients older than 18 years, admitted to ICU for respiratory distress due to community- acquired pneumonia , with a microbiologically confirmed absence of influenza (for inclusion in the control group)

Exclusion Criteria:

* Age < 18 years old
* Pregnant women
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill community-acquired pneumonia patients
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2019-01-18 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Difference in immune cell profile in blood between influenza and non-influenza CAPIV patients at ICU. | through study completion, after 3 influenza seasons (3 years)
  Immunophenotyping of blood will be performed to determine number of neutrophils, T- and B-cell subsets, NK cell and myeloid cell subsets. Difference in influenza positive and influenza negative patients is expected.
Difference in cytokine production of mononuclear cells to fungal stimulation in blood between influenza and non-influenza CAPIV patients at ICU. | through study completion, after 3 influenza seasons (3 years)
  Key cytokine reaction of mononuclear cells (PBMC) after fungal stimulation will be performed. Difference in influenza positive and influenza negative patients is expected.
Difference in function of blood neutrophils between influenza and non-influenza CAPIV patients at ICU. | through study completion, after 3 influenza seasons (3 years)
  Functional analysis by killing assay will be performed.
Difference in in immune cell profile in BAL fluid between influenza and non-influenza CAPIV patients at ICU. | through study completion, after 3 influenza seasons (3 years)
  Immunophenotyping of BAL fluid will be performed to determine number of neutrophils, T- and B-cell subsets, NK cell and myeloid cell subsets. Difference in influenza positive and influenza negative patients is expected.
Difference in cytokine production of mononuclear cells to fungal stimulation in BAL fluid between influenza and non-influenza CAPIV patients at ICU. | through study completion, after 3 influenza seasons (3 years)
  Key cytokine reaction of mononuclear BAL fluid cells after fungal stimulation will be performed. Difference in influenza positive and influenza negative patients is expected.
Difference in function of BAL fluid neutrophils between influenza and non-influenza CAPIV patients at ICU. | through study completion, after 3 influenza seasons (3 years)
  Functional analysis by killing assay will be performed.
Difference in pathological hallmarks between influenza and non-influenza CAPIV patients at ICU. | through study completion, after 3 influenza seasons (3 years)
  Biopsies of respiratory tract tissue will be compared between two groups.

SECONDARY OUTCOMES:
Difference in longitudinal alterations in phagocytic cell and mononuclear inflammatory cell subsets in blood and BAL fluid and their response to fungal stimulation between the main study arms. | through study completion, after 3 influenza seasons (3 years)
  Longitudinal alterations in advanced immunophenotyping results and (fungal) cell stimulation will be analysed and compared between groups.
Longitudinal differences in anatomopathological characteristics of the respiratory tract in CAPIV +/- influenza | through study completion, after 3 influenza seasons (3 years)
  Respiratory tract biopsies will be compared longitudinally throughout the disease course.
Correlation of findings with invasive pulmonary aspergillosis incidence | through study completion, after 3 influenza seasons (3 years)
  All data will be compared within each group between patients that develop IPA vs no development of IPA.
Correlation of findings with outcome | through study completion, after 3 influenza seasons (3 years)
  All data will be compared to outcome measures (length of ICU stay, mortality, etc) to find hallmarks of severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Joost Wauters, PhD, Principal Investigator — UZ Leuven
Locations (1):
- Universitaire Ziekenhuizen Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided